CLINICAL TRIAL: NCT06239012
Title: SAPA Study (Seated Posture Analysis System) : Reliability and Validity Evaluation of the BePoW Device
Brief Title: Reliability and Validity Evaluation of the BePoW Device
Acronym: SAPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pôle Saint Hélier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-A00609-36
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Position Sense Disorders
MeSH Terms: conditions — Somatosensory Disorders

STUDY DESIGN:
Intervention Model Description: exploratory, monocentric, reliability-validity clinical investigation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- position measurement with BePoW device compared with MCPAA scale measurements (Experimental): Each patient will have position measurement with BePoW device and, at the same time, will have MCPAA scale measurements
  Interventions: Device: Position measurement with BePow; Other: Position measurement with MCPAA scale

INTERVENTIONS:
Device: Position measurement with BePow — 14 measurements taken with the device
Other: Position measurement with MCPAA scale — MCPAA : measurement of seated postural control in adults in French 12 measurements taken with the goniometer

SUMMARY:
The aim of this clinical investigation is to develop a reliable and valid device to instantly measure the subject's sitting posture in a wheelchair, without using the MCPAA scale.

DETAILED DESCRIPTION:
Each subject will be invited to a single experimental session lasting approximately one hour, during which all assessments will be performed.

During the visit, the patient will complete an autonomy questionnaire and assess wheelchair fatigue. A spirometry test will be performed.

The measurements will then be recorded by the BePoW software and the occupational therapist.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age,
* Having freely consented to participate in the study (or their legal representative in the case of guardianship, in agreement with the patient),
* In the case of a guardianship, the legal representative having read the information document intended for the legal guardian of an adult under legal protection (under guardianship) and given his/her free and informed consent for the person for whom he/she is responsible to participate in the study (in agreement with the patient).
* Temporarily or permanently wheelchair-bound,
* Affiliated with a social security scheme or beneficiary of such a scheme.

Exclusion Criteria:

* Has comprehension problems that prevent him/her from giving free and informed consent and from completing the investigation (following instructions, answering questionnaires),
* Suffering from a pathology (Huntington's disease, Sydenham's Chorea) preventing stable sitting posture during participation in the investigation,
* Have undergone an amputation that prevents the BePoW device from taking measurements,
* having undergone a tracheotomy preventing spirometry.
* Pregnant, parturient or breast-feeding women,
* Person deprived of liberty by a judicial decision (except guardianship or curatorship) or or administrative decision, a person under psychiatric care or admitted to a or social establishment for purposes other than research,
* Minors,
* Person in an emergency situation unable to give prior consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-02-29 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
Reliability assessment: intraclass correlation coefficient (ICC) between BePoW measurements | Immediately after inclusion
  12 data records for each measurement for intra ICC
Validity assessment: correlation coefficient r between raw goniometric measurements and BePoW measurements, | Immediately after inclusion
  kappa coefficient between recoded measurements : BePow / MCPAA

SECONDARY OUTCOMES:
Assess the validity of BePoW measurements in relation to fatigability. | Immediately after inclusion
  assessment using a visual numerical scale, from 0 to 10
Assess the validity of BePoW measurements in relation to autonomy. | Immediately after inclusion
  assessment by the MIF (Measure of Functional Independence) questionnaire from 21 (total dependence) to 47 (completely independent)
Assessing the validity of BePoW measurements in relation to respiratory capacity | Immediately after inclusion
  assessed by the ratio of forced expiratory volume in one second (FEV1) to FEV1 at 6 seconds (FEV 6).
  Spirometry will be performed 3 times, with the highest value retained.
Determine the standard error measurement (SEM) on angular measurements taken by BePoW | Immediately after inclusion
  Calculation of the standard error measurement (SEM) of each measurement taken by the device.
Determining the minimum detectable change (MDC) on angular measurements taken by BePoW | Immediately after inclusion
  Calculation of the minimum detectable change (MDC) of each measurement taken by the device.

CONTACTS AND LOCATIONS:
Locations (1):
- Pôle Saint Hélier, Rennes, Brittany Region, France